CLINICAL TRIAL: NCT05309291
Title: A Randomized, Open-label, Controlled, Parallel, Multicenter Study in Kidney Failure Patients on Hemodialysis Comparing the Theranova Dialyzer to Hemodiafiltration
Brief Title: Theranova Randomized, Controlled, Trial (RCT) in China
Acronym: ROCKet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vantive Health LLC (Industry)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BXU561424
Record Dates: First submitted 2022-03-25; First posted 2022-04-04 (Actual); Results first posted 2024-10-15 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Chronic Kidney Failure; Acute Kidney Failure
MeSH Terms: conditions — Kidney Failure, Chronic; Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Theranova 400 Dialyzer (Experimental): 1 week, 1 session in mid-week HD therapy. Pre dialysis blood samples taken from fistula needle or central venous catheter. Post dialysis blood samples taken from arterial sampling port of bloodline
  Interventions: Device: Theranova 400 Dialyzer
- FX 800 Dialyzer (Active Comparator): 1 week, 1 session in mid-week HDF therapy. Pre dialysis blood samples taken from fistula needle or central venous catheter. Post dialysis blood samples taken from arterial sampling port of bloodline
  Interventions: Device: FX 800 Dialyzer

INTERVENTIONS:
Device: Theranova 400 Dialyzer — Dialysis performed in HD mode.
  Other Names: Hollow fiber dialyzers with medium cut-off membrane
  Arms: Theranova 400 Dialyzer
Device: FX 800 Dialyzer — Dialysis performed in HDF mode.
  Other Names: Hollow fiber hemodialysis filter
  Arms: FX 800 Dialyzer

SUMMARY:
Traditional hemodialysis (HD) therapy is very effective in clearing urea and smaller middle molecules, but is limited in clearing larger middle molecules. These accumulated large middle-molecular-weight uremic toxins may cause and aggravate inflammation, atherosclerosis and calcification, which can indirectly lead to the death of patients. Studies have shown that, compared to conventional high-flux HD (HF-HD), hemodiafiltration (HDF) that combines diffusion and convection can reduce the all-cause mortality. Compared to the conventional HF-HD, HDF can more effectively clear larger molecular toxins in one session, which may be related to the better clearance effect of HDF on middle-molecular-weight toxins

Theranova's innovative Medium Cut-Off® membranes has high permeability and selectivity to uremic toxins (clearance of a molecular weight of up to 45 kDa) and can retain essential proteins, to maintain patient's albumin level during the HD treatment[9]. Its unique membrane and high cut-off characteristics expand the clearance range beyond those of flux membrane dialyzers. Theranova 400 can be widely used in most blood purification centers under conventional HD equipment and treatment modes, with the effect similar to HDF This study is to demonstrate non-inferiority of the Theranova 400 Dialyzer in HD mode (hereinafter referred to as Theranova 400) compared to HDF, using FX 800 in HDF mode (hereinafter referred to as FX 800).

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥18 years old and ≤80 years old, regardless of gender;
2. Patients who are able to sign informed consent form (ICF) after an explanation of the proposed study;
3. Patients who receive in-center HD treatment at a site that routinely implements high flux dialysis and HDF;
4. Patients who have been stable receiving in-center HD/HDF for >3 months prior to study enrollment;
5. Patients with kidney failure receiving maintained HD treatment with a history of thrice weekly HD, and at least 1 HDF session within 1 month prior to the study shall be judged by the investigator;
6. Patients who have an adequate arteriovenous (AV) fistula or graft, or dual-lumen tunneled catheter capable of providing a blood flow rate (QB) of at least 250 mL/min;
7. Patients have no changes in dialysis prescription (dialyzer, time, dialysis fluid flow rate (QD), QB, sufficient dialysis anticoagulation, and stable prescribed doses) over last 6 treatments as judged by the investigator. The dialysis treatment time should be 3.5 to 4.5 hours per session with minimum QB of 250 mL/min and QD of 500 mL/min;
8. Patients with a minimum total convective volume (including ultrafiltration (UF)) of 16 L post-dilution for the most recent HDF treatment;
9. Patients who have Kt/Vurea > 1.2 for the last 2 measurements, with the most recent Kt/Vurea measurement taken within 4 weeks before or during study screening.

Exclusion Criteria:

1. Patients who have acute kidney injury with the chance for recovery;
2. Pregnant and lactating women;
3. Patients diagnosed with a New York Heart Association (NYHA) Class IV congestive heart failure, or acute coronary syndrome, and/or who have suffered a myocardial infarction within 3 months prior to the start of the study;
4. Patients with known hemodynamic instability, anemia (hemoglobin <90 g/L), and/or patients with hemoglobin >130g/L for coagulation risk;
5. Patients with active or ongoing infection as per investigator's judgement (e.g C-reactive protein [CRP] level more than 5 folds of normal);
6. Patients who are severely malnourished or with significant disease that interferes with liver synthetic function ( e.g. with serum albumin <30 g/L);
7. Patients with positive serology tests for Hepatitis B surface antigen, Hepatitis C total antibody, and advanced liver, or pulmonary disease as judged by the investigator;
8. Patients with positive serology tests for human immunodeficiency virus (HIV), Syphilis;
9. Patients receiving immunosuppressive treatment or with autoimmune disease;
10. Patients with a history of solid tumors requiring anti-cancer therapy in the past or next 6 months, or with a life expectancy of <1 year, or patients with history of hematology neoplasm;
11. Patients who are pre-scheduled for a living donor kidney transplant within the next 1 year, who plan a change to peritoneal dialysis (PD) within the next 1 year, or who require single-needle dialysis therapy;
12. Patients who have had an allergic response to polyarylethersulfone (PAES) or polysulfone (PS) membrane or have history of poor tolerance to dialyzers with synthetic membranes;
13. Patients with a history of severe mental disorders who are unable to provide consent or comply with study procedures as assessed by the investigator;
14. Patients who are currently participating in or have previously participated in other interventional clinical studies during the past 30 days;
15. Patients with any comorbidity possibly conflicting with the study as judged by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 323 (Actual)
Dates: Start 2022-06-22 (Actual); Primary Completion 2023-07-06 (Actual); Study Completion 2023-07-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - Investigational Site, Beijing
  - Investigational Site, Dalian
  - Investigational Site, Hangzhou
  - Investigational Site, Nanjing
  - Investigational Site, Shanghai
  - Investigational Site, Shenzhen
  - Investigational Site, Suzhou

IPD SHARING:
Plan to Share IPD: Yes
Sharing of Clinical Trial Data: Sponsor is committed to sharing clinical trial data with external medical experts and scientific researchers in the interest of advancing public health. As such, the Sponsor will supply anonymized Individual Patient Datasets (IPD) and supporting documents (synopsis of clinical study reports, protocol and SAP's)
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Upon approval of a legitimate research request.
Access Criteria: Research requests will be reviewed by qualified medical and scientific experts within the company. If the Sponsor agrees to the release of clinical data for research purposes, the requestor will be required to sign a data sharing agreement (DSA) in order to ensure protection of patient confidentiality and any intellectual property rights of the Sponsor prior to the release of any data.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited across 11 investigational sites in China, between June 2022 and July 2023.
Pre-assignment Details: Of the 323 patients enrolled, 274 patients met the study entry criteria and were randomized for treatment.
Groups:
- Theranova 400 Dialyzer: 1 week, 1 mid-week HD therapy session.
  Theranova 400 Dialyzer: Dialysis performed in HD mode.
- FX 800 Dialyzer: 1 week, 1 mid-week HDF therapy session.
  FX 800 Dialyzer: Dialysis performed in HDF mode.
Period: Overall Study
Arm/Group | Theranova 400 Dialyzer | FX 800 Dialyzer
Started | 138 | 136
As Treated (All enrolled patients who were treated; based on actual treatment received. Note: 1 patient was treated with the incorrect device after randomization, (i.e., the patient was assigned to the FX800 group according to randomization result but was treated with Theranova 400).) | 139 | 135
Completed | 138 | 135
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Theranova 400 Dialyzer | FX 800 Dialyzer | Total
Number analyzed (Participants) | 138 | 136 | 274
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.1 (11.99) | 53.0 (11.43) | 52.6 (11.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 35 | 79
  Male | 94 | 101 | 195
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Chinese | 138 | 135 | 273
  Ethnicity: Unknown | 0 | 1 | 1
Child-bearing potential [Count of Participants; unit: Participants] — Population: Child-bearing potential outcome measure was assessed only in female participants
  Participants
    Yes: number analyzed (Participants) | 44 | 35 | 79
    Yes | 15 | 12 | 27
    No: number analyzed (Participants) | 44 | 35 | 79
    No | 29 | 23 | 52
Dialysis Vintage [Mean (Standard Deviation); unit: years] | 7.17 (4.86) | 6.28 (4.45) | 6.73 (4.67)
Weight [Mean (Standard Deviation); unit: kg] | 65.00 (10.62) | 66.39 (11.15) | 65.69 (10.89)
Dry Weight [Mean (Standard Deviation); unit: kg] | 62.47 (10.39) | 63.97 (10.97) | 63.22 (10.69)
Height [Mean (Standard Deviation); unit: cm] | 167.86 (7.28) | 168.92 (7.58) | 168.39 (7.44)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 23.02 (3.17) | 23.20 (3.19) | 23.11 (3.17)

OUTCOME MEASURES:

1. Primary Outcome: Reduction Ratio (RR) of Lambda Free Light Chains (λ FLC)
Description: One mid-week treatment day dialysis session, pre-dialysis and post-dialysis. The RR was calculated using the following formula:
  [(Cpre-Cpost)/Cpre], where Cpre and Cpost were the arterial plasma concentrations of λ FLC measured pre- and post- the mid-week dialysis session, respectively
Time Frame: Assessed at the mid-week treatment day dialysis session
Population: The per-protocol set (PPS) is a subset of patients who were randomized to the respective treatment at the mid-week treatment day dialysis session and did not have any major protocol deviations that could affect the assessment of the primary endpoint.
Measure: Mean (95% Confidence Interval); unit: Reduction Ratio (%)
Groups:
- Theranova 400 Dialyzer: 1 week, 1 mid-week HD therapy session .
  Theranova 400 Dialyzer: Dialysis performed in HD mode.
Arm/Group | Theranova 400 Dialyzer | FX 800 Dialyzer
Number analyzed (Participants) | 131 | 131
Reduction Ratio (%) | 36.02 [34.36 to 37.69] | 19.03 [17.64 to 20.41]
Statistical Analysis 1: Comparison: Theranova 400 Dialyzer vs FX 800 Dialyzer; Non-inferiority of the Theranova 400 Dialyzer compared to the FX 800 Dialyzer in regard to the λ FLC RR at the mid-week treatment day dialysis session was assessed; Test type: Non-Inferiority — The null hypothesis to demonstrate non-inferiority using a 10% margin for λ FLC RR can be expressed as: Ho: μT-μR ≤ -3.783. The alternative hypothesis is expressed as: Ha: μT-μR > -3.783 where μT denotes the Theranova 400 treatment mean and μR denotes the FX 800 treatment mean; p < 0.0001, t-test, 2 sided; T-test was utilized to generate a two-sided 95% confidence interval (CI) for the difference in means; Mean Difference (Final Values) = 16.99, 95% CI 2-sided [14.84 to 19.15], Standard Deviation 8.86

2. Primary Outcome: Reduction Ratio of Beta-2 Microglobulin (β2-MG)
Description: One mid-week treatment day dialysis session, pre-dialysis and post-dialysis. The RR was calculated using the following formula:
  [(Cpre-Cpost)/Cpre], where Cpre and Cpost were the arterial plasma β2-MG concentrations measured pre- and post- the mid-week dialysis session, respectively.
Time Frame: Assessed at the mid-week treatment day dialysis session
Population: The per-protocol set (PPS) was a subset of patients who were randomized to the respective treatment at the mid-week treatment day dialysis session and did not have any major protocol deviations that could affect the assessment of the primary endpoint.
Measure: Mean (95% Confidence Interval); unit: Reduction Ratio (%)
Arm/Group | Theranova 400 Dialyzer | FX 800 Dialyzer
Number analyzed (Participants) | 131 | 131
Reduction Ratio (%) | 77.03 [76.15 to 77.91] | 78.22 [77.18 to 79.25]
Statistical Analysis 1: Comparison: Theranova 400 Dialyzer vs FX 800 Dialyzer; Non-inferiority of the Theranova 400 Dialyzer compared to the FX 800 Dialyzer in regard to the β2-MG RR at the mid-week treatment day dialysis session was assessed; Test type: Non-Inferiority — The null hypothesis to demonstrate non-inferiority using a 10% margin for ß2-MG RR can be expressed as Ho: μT-μR ≤ -7.848. The alternative hypothesis is expressed as: Ha: μT-μR > -7.848, where μT denotes the Theranova 400 treatment mean and μR denotes the FX 800 treatment mean; p < 0.0001, t-test, 2 sided; T-test was utilized to generate a two-sided 95% confidence interval (CI) for the difference in means; Mean Difference (Final Values) = -1.19, 95% CI 2-sided [-2.54 to 0.16], Standard Deviation 5.55

ADVERSE EVENTS:
Time Frame: All treatment emergent adverse events collected from enrollment through the End of Study Visit, i.e., a follow-up visit during the end-of-week dialysis session (up to 1 week)
Description: The safety analysis set included all enrolled patients, as treated (139 patients in the Theranova 400 group and 135 patients in the FX 800 group)
Arm/Group | Theranova 400 Dialyzer | FX 800 Dialyzer
All-Cause Mortality (participants affected / at risk) | 0/139 | 0/135
Serious Adverse Events (participants affected / at risk) | 1/139 | 0/135
Other Adverse Events (participants affected / at risk) | 0/139 | 0/135
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Theranova 400 Dialyzer (N=139) | FX 800 Dialyzer (N=135)
Arteriovenous fistula occlusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Baxter Healthcare Corporation reserves the right of prior review and approval of data from this study relative to the potential release of proprietary information to any publication or for any presentation.

DOCUMENTS (2):
  • Study Protocol (2022-05-30): https://cdn.clinicaltrials.gov/large-docs/91/NCT05309291/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-28): https://cdn.clinicaltrials.gov/large-docs/91/NCT05309291/SAP_001.pdf